CLINICAL TRIAL: NCT04798183
Title: Geometrical Facial Deformation According to Posture and Non-invasive Ventilation Mask Virtual Fit in Amyotrophic Lateral Sclerosis
Brief Title: Geometrical Facial Deformation According to Posture in Amyotrophic Lateral Sclerosis
Status: Completed | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sungchul Huh, Medical doctor, Pusan National University Yangsan Hospital
Other Study IDs: 05-2021-034
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy participants: A healthy person with no history of facial surgery or paralysis.
  Interventions: Diagnostic Test: 3-dimensional scan
- Amyotrophic Lateral Sclerosis with bulbar involvement patients: Amyotrophic lateral sclerosis with no history of facial surgery or paralysis
  Interventions: Diagnostic Test: 3-dimensional scan

INTERVENTIONS:
Diagnostic Test: 3-dimensional scan — Facial 3-dimensional scan according to posture

SUMMARY:
The measurement of the facial deformation according to the body posture will be conducted by 3D scanning for each posture after marking the landmarks on the face. A 3D scan of the face will be conducted for 1 minute in a static state for the sitting posture to be used as a reference, the supine posture to gaze at the ceiling while lying down correctly, and the lateral posture to the side with the upper body facing left. Healthy volunteer and ALS with bulbar palsy participants will be asked to keep their mouths closed gently while the 3D scan was being processed. A post-processing of the 3D face scan data will be conducted to analyze facial deformation by the body postures. A facial deformation will be analyzed by measuring the amount of change in position for each reference point after aligning and rotating the facial data on the same basis. The relative ratio of the amount of position change to the size of the face will be analyzed. The present study will analyze the effect of the body posture on the position changes of the landmarks.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a progressive neurodegenerative disease that eventually affects the respiratory muscles. In most cases of the slow progression of respiratory failure, noninvasive ventilation (NIV) is the first treatment option. NIV treatment provides a better quality of life and is, therefore, strongly recommended; however, its use must consider the type of ALS. Severe bulbar dysfunction limits NIV treatment. Aside from additional NIV options in ALS, including mouthpiece ventilation and intermittent abdominal pressure ventilation, prolonged use of a ready-made face mask is impractical for several reasons. Cognitive impairments can affect the maintenance of NIV. Hypersalivation and bronchial secretion disrupting ventilation can lead to poor NIV adherence. Pressure injuries are another clinical issue. The incidence of pressure injuries associated with NIV masks ranges from 10-31%. Long-term use of NIV face masks can result in pressure injuries at the contact area, and skin-protective patches may not prevent skin problems. Patients with bulbar ALS frequently have postural facial deformations, and these can lead to difficulties in wearing the NIV mask.

The aim of this study was to compare the deformations of the face in different postures in subjects with bulbar ALS and healthy participants. This study also virtually fitted an NIV mask to understand how the NIV mask interface affects the face in different postures.

ELIGIBILITY:
Inclusion Criteria:

1. Patient

   * a patient with Amyotrophic Lateral Sclerosis over 16 years
   * a patient with respiratory difficulty
   * a patient who requires or anticipates mechanical ventilation
   * a patient who visit out- or inpatient clinic at rehabilitation hospital
2. Healthy volunteer

   * a volunteer without history of facial surgery or neuromuscular disease
   * a volunteer without respiratory difficulty

Exclusion Criteria:

1. Patient

   * a patient who cannot scan due to respiratory instability
   * a patient who cannot bear posture for 3D scanning
2. Healthy volunteer

   * a volunteer with neuromuscular disease
   * a volunteer with history of facial surgery or palsy

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patient: a patient who visit out- or inpatient clinic at rehabilitation hospital Healthy volunteer: community dwelling volunteer
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Yeon Kim, PhD, Study Director — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Participants | Amyotrophic Lateral Sclerosis With Bulbar Involvement Patients
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of people enrolled in the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Participants | Amyotrophic Lateral Sclerosis With Bulbar Involvement Patients | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (9.2) | 41 (8.8) | 40.5 (9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex/Gender was not collected from any participants because it was not a major variable influencing the result value
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: The Amounts of Change of Landmarks Position According to Posture
Description: The primary outcome measure is the change in position of anatomical landmarks, quantified using millimeter measurements in the anteroposterior and lateral directions. Change is reported as the mean displacement (mm) during the change in position from the initial position (sitting) to the subsequent position (supine & side-lying). Ten anatomical landmarks were located in the nasal root area for 4 points (sellion, glabella, left dacryon, and right dacryon) and in the oral area for 6 points (subnasale, SN; labial superius, LS; labial inferius, LI; cheilion left, CL; cheilion right, CR; and promentale, PM)
Time Frame: 1 minute
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Bulbar ALS: Amyotrophic Lateral Sclerosis with bulbar involvement patients
Arm/Group | Healthy Participants | Bulbar ALS
Number analyzed (Participants) | 14 | 14
mm
  movement of landmarks according to postural change from sitting to supine | 1.0 (0.9) | 2.4 (2.2)
  movement of landmarks according to postural change from sitting to lateral decubitus | 2.9 (1.4) | 5.6 (3.2)

ADVERSE EVENTS:
Time Frame: Adverse events are observed from the time of study enrollment until all procedures are performed and outcome measures are measured. Participants usually complete all procedures within 1 day.
Arm/Group | Healthy Participants | Bulbar ALS
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

LIMITATIONS AND CAVEATS:
The face in a real situation with the NIV strap may differ from that in the virtual simulation without the NIV strap. Wearing an NIV mask could alleviate the effect of facial deformation caused by posture, but 3-dimensional scanning could not be accomplished while wearing a mask.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT04798183/Prot_SAP_000.pdf